CLINICAL TRIAL: NCT04707339
Title: Management of Acute Appendicitis at District General Hospital
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Princess Alexandra Hospital NHS Trust (Other)
Responsible Party: Principal Investigator, Naveed Kirmani, Principal Investigator, Princess Alexandra Hospital NHS Trust
Other Study IDs: 3810
Record Dates: First submitted 2021-01-11; First posted 2021-01-13 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Appendicitis Acute; Covid19
Keywords: Acute Appendicitis; COVID-19 pandemic; Management
MeSH Terms: conditions — Appendicitis; COVID-19 | interventions — Appendectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acute Appendicitis pre-COVID management: Audit of Acute appendicitis management in 2017-18
  Interventions: Procedure: Appendicectomy
- Acute Appendicitis during COVID management: Audit of Acute appendicitis management in 2020
  Interventions: Procedure: Appendicectomy

INTERVENTIONS:
Procedure: Appendicectomy — Laparoscopic or Open Appendicectomy

SUMMARY:
The Investigators aim to assess;

1. whether the changes in managing patients during COVID has reduced the negative appendicectomy rate?
2. compare the difference in outcomes of conservatively and surgically managed Acute Appendicitis?
3. Whether there uniformity in prescribing postoperative antibiotics with resultant outcomes?
4. Whether the incidence of complicated appendicitis has increased?

DETAILED DESCRIPTION:
As acute appendicitis is the most commonly managed emergency presentation for surgeons, the investigators aim to assess whether the changes in managing patients during COVID has reduced the negative appendicectomy rate, to compare the difference in outcomes of conservatively and surgically managed Acute Appendicitis? to assess whether there uniformity in prescribing postoperative antibiotics with resultant outcomes? to assess whether the incidence of complicated appendicitis has increased? This will be a single centre retrospective observational study. All the patients presenting in A&E department with a diagnosis of acute appendicitis to be included. the only exclusion criteria are the age of participants for less than 5 years. The data will be analysed and calculated using SPSS version 23.

ELIGIBILITY:
Inclusion Criteria:

* All participants reporting in accident and emergency with a diagnosis of acute appendicitis irrespective of age above 5 years, gender and morbidities (this group for conservative management)

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients with a diagnosis of Acute Appendicitis will be included
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-01-30 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2021-01-30 (Estimated)

PRIMARY OUTCOMES:
Negative Appendicectomy Rate | 8 months
  Negative appendicectomy rate will be calculated to define the benefits of increasing the preoperative scanning in the form of ultrasound, CT scan or both.
Outcomes of Conservative vs Operative Management | 8 months
  The outcomes of both conservatively and operatively managed patients will be assessed to define the best management approach.
Increased Open Appendicectomy Rate | 8 months
  The rate of laparoscopic to open and open appendicectomy rate will be calculated to understand if the surgical practice has been changed during COVID-19 pandemic?
Surgical site infection in patients on antibiotics | 8 months
  The rate of incidence of superficial and deep wound infection will be calculated to define the applicability of use of Antibiotics

SECONDARY OUTCOMES:
Length of Stay | 8 months
  The number of days of postoperative admission in hospital will be assessed while comparing the type of surgery and co-morbidities.

CONTACTS AND LOCATIONS:
Overall Officials: Naveed Kirmani, FRCS, Principal Investigator — The Princess Alexandra Hospital NHS Trust
Locations (1):
- The Princess Alexandra Hospital NHS Trust, Harlow, Essex, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hori T, Machimoto T, Kadokawa Y, Hata T, Ito T, Kato S, Yasukawa D, Aisu Y, Kimura Y, Sasaki M, Takamatsu Y, Kitano T, Hisamori S, Yoshimura T. Laparoscopic appendectomy for acute appendicitis: How to discourage surgeons using inadequate therapy. World J Gastroenterol. 2017 Aug 28;23(32):5849-5859. doi: 10.3748/wjg.v23.i32.5849. PMID 28932077
- [Background] van den Boom AL, de Wijkerslooth EML, van Rosmalen J, Beverdam FH, Boerma EG, Boermeester MA, Bosmans JWAM, Burghgraef TA, Consten ECJ, Dawson I, Dekker JWT, Emous M, van Geloven AAW, Go PMNYH, Heijnen LA, Huisman SA, Jean Pierre D, de Jonge J, Kloeze JH, Koopmanschap MA, Langeveld HR, Luyer MDP, Melles DC, Mouton JW, van der Ploeg APT, Poelmann FB, Ponten JEH, van Rossem CC, Schreurs WH, Shapiro J, Steenvoorde P, Toorenvliet BR, Verhelst J, Versteegh HP, Wijnen RMH, Wijnhoven BPL. Two versus five days of antibiotics after appendectomy for complex acute appendicitis (APPIC): study protocol for a randomized controlled trial. Trials. 2018 May 2;19(1):263. doi: 10.1186/s13063-018-2629-0. PMID 29720238
- [Background] Ferguson DM, Parker TD, Arshad SA, Garcia EI, Hebballi NB, Tsao K. Standardized Discharge Antibiotics May Reduce Readmissions in Pediatric Perforated Appendicitis. J Surg Res. 2020 Nov;255:388-395. doi: 10.1016/j.jss.2020.05.086. Epub 2020 Jun 29. PMID 32615311
- [Background] Javanmard-Emamghissi H, Boyd-Carson H, Hollyman M, Doleman B, Adiamah A, Lund JN, Clifford R, Dickerson L, Richards S, Pearce L, Cornish J, Hare S, Lockwood S, Moug SJ, Tierney GM; COVID: HAREM (Had Appendicitis, Resolved/Recurred Emergency Morbidity/Mortality) Collaborators Group. The management of adult appendicitis during the COVID-19 pandemic: an interim analysis of a UK cohort study. Tech Coloproctol. 2021 Apr;25(4):401-411. doi: 10.1007/s10151-020-02297-4. Epub 2020 Jul 15. PMID 32671661
- [Background] RIFT Study Group on behalf of the West Midlands Research Collaborative. Appendicitis risk prediction models in children presenting with right iliac fossa pain (RIFT study): a prospective, multicentre validation study. Lancet Child Adolesc Health. 2020 Apr;4(4):271-280. doi: 10.1016/S2352-4642(20)30006-7. Epub 2020 Feb 13. PMID 32200936